CLINICAL TRIAL: NCT03210298
Title: Multicenter, International Online Documentation of Indications and Results of Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC Und PITAC) for Treating Malignant Peritoneal and Pleural Diseases
Brief Title: International Registry of Patients Treated With Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC)
Acronym: PIPACRegis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sabine Rhode (Other)
Collaborators: Ruhr University of Bochum (Other)
Responsible Party: Sponsor-Investigator, Sabine Rhode, Coordinator, University of Magdeburg
Organization: University of Magdeburg (Other)
Other Study IDs: RUB 15-5280
Record Dates: First submitted 2017-06-29; First posted 2017-07-06 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Peritoneum Cancer; Peritoneum Neoplasm; Pleural Cancer; Pleural Effusion; Pleural Mesothelioma; Ovarian Cancer; Gastric Cancer; Appendix Cancer; Pseudomyxoma Peritonei; Colorectal Cancer; Pancreas Cancer; Gallbladder Cancer; Ascites; CUP; Chemotherapeutic Toxicity
Keywords: Pressurized IntraPeritoneal Aerosol Chemotherapy; PIPAC; Pressurized IntraThoracic Aerosol Chemotherapy; PITAC; Cisplatin; Oxaliplatin; Gemcitabine; Paclitaxel; nab-Paclitaxel; Doxorubicine; Mitomycin
MeSH Terms: conditions — Peritoneal Neoplasms; Pleural Effusion; Mesothelioma, Malignant; Ovarian Neoplasms; Stomach Neoplasms; Appendiceal Neoplasms; Pseudomyxoma Peritonei; Colorectal Neoplasms; Pancreatic Neoplasms; Gallbladder Neoplasms; Ascites | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Peritoneal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Combination Product: PIPAC — A chemotherapeutic solution is aerosolized into the expanded abdominal cavity during laparoscopy, under pressure. This allows a relatively homogeneous repartition of the drug and an effective tissue penetration.
  Other Names: PITAC; Intraperitoneal chemotherapy; Intrathoracic chemotherapy

SUMMARY:
Multicentric, international, web-based prospective documentation of the indications and results of Pressurized Aerosol Chemotherapy (so-called PIPAC or PITAC) for treating malignant pleural and peritoneal diseases. Indication is decided by the treating physician. There are no predefined inclusion or exclusion criteria.

DETAILED DESCRIPTION:
All data entered into the registry documenting the patient cohort characteristics (disease, demography, therapy) are analyzed using descriptive statistics. Survival data are analyzed with Kaplan-Meier statistics. Multivariate Cox Proportional Hazard Models are used to identify potential prognostic and predictive factors. In particular, a risk- adjusted comparison of the outcome criteria with a propensity score is planned.

The data are stored in a SQL-based online database. Patient data are pseudoanonymized. The registry has received approval of the data protection officer of the State of Northrhine-Westphalia.

The study steering committee is blinded towards the identity of the participating institutions. Each participating institution receives an annual report with own data vs. benchmark. Scientific analysis can be proposed by the steering committee, by a participating institution or by other scientists, subjected to the approval of the independent scientific advisory board.

An export function has been built in to allow data exchange with the HIPEC Registry of the German Society for General and GI surgery (http://www.dgav.de/studoq/studoqhipec.html).

ELIGIBILITY:
Inclusion criteria:

* verified peritoneal metastasis
* colorectal cancer
* ovarian cancer
* gastric cancer
* appendical cancer
* pseudomyxoma peritonei
* malignant mesothelioma
* pancreatic cancer
* gallbladder cancer
* small bowel cancer

Exclusion criteria

- bowel obstruction

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In the rule, pretreated patients with chemoresistant peritoneal metastasis of various origins.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 to 5 years
  Kaplan-Meier

SECONDARY OUTCOMES:
Clinical Benefit Rate | 3 months
  according to RECIST criteria (CR + PR + SD)
Histological tumor regression according to the Peritoneal Regression Grading Score (PRGS) | 6 weeks
  according to the Peritoneal Regression Grading Score (PRGS)
Safety according to CTCAE 4.0 | 6 weeks
  according to CTCAE 4.0
Quality of life according to QLQ-30 of EORTC | 6-18 weeks
  according to QLQ-30 of EORTC

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Horvath, MD, Principal Investigator — University Hospital Tuebingen
Locations (16):
- Roffo Cancer Institute, Buenos Aires, Argentina
- Peter MacCallum Cancer Centre, Melbourne, Australia
- SALK - Salzburger Landeskliniken, Salzburg, Austria
- University Hospital Gent (UZ Gent), Ghent, Belgium
- University Hospital Odense, Odense, Denmark
- France (4):
  - Centre Hospitalier Universitaire, Grenoble
  - Centre Hospitalier Universitaire, Lille
  - Hospices civils de Lyon, Lyon
  - Centre du Cancer, Montpellier
- University Hospital Tübingen, Tübingen, Germany
- IRCC Torino Candiolo, Turin, Italy
- F. Łukaszczyk Oncology Centre, Bydgoszcz, Poland
- Gersten Institute for Cancer Research, Moscow, Russia
- National University Hospital, Singapore, Singapore
- Hospital de Pilar, Barcelona, Spain
- University Hospital Lausanne CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Requests can be addressed to the Scientific Advisory Board, AnInstitut für Qualitässicherung in der operativen Medizin gGmbH, Leipziger Str. 44, 39120 MAGDEBURG, Germany
Supporting Information: Study Protocol, ICF
Time Frame: until 2021/12/31
Access Criteria: Approval through the independent scientific advisory board of the Institut for Quality Control, see above

REFERENCES:
- [Background] Graversen M, Detlefsen S, Bjerregaard JK, Pfeiffer P, Mortensen MB. Peritoneal metastasis from pancreatic cancer treated with pressurized intraperitoneal aerosol chemotherapy (PIPAC). Clin Exp Metastasis. 2017 Jun;34(5):309-314. doi: 10.1007/s10585-017-9849-7. Epub 2017 May 17. PMID 28516306
- [Background] Grass F, Vuagniaux A, Teixeira-Farinha H, Lehmann K, Demartines N, Hubner M. Systematic review of pressurized intraperitoneal aerosol chemotherapy for the treatment of advanced peritoneal carcinomatosis. Br J Surg. 2017 May;104(6):669-678. doi: 10.1002/bjs.10521. PMID 28407227
- [Background] Hubner M, Teixeira Farinha H, Grass F, Wolfer A, Mathevet P, Hahnloser D, Demartines N. Feasibility and Safety of Pressurized Intraperitoneal Aerosol Chemotherapy for Peritoneal Carcinomatosis: A Retrospective Cohort Study. Gastroenterol Res Pract. 2017;2017:6852749. doi: 10.1155/2017/6852749. Epub 2017 Feb 26. PMID 28331493
- [Background] Teixeira Farinha H, Grass F, Kefleyesus A, Achtari C, Romain B, Montemurro M, Demartines N, Hubner M. Impact of Pressurized Intraperitoneal Aerosol Chemotherapy on Quality of Life and Symptoms in Patients with Peritoneal Carcinomatosis: A Retrospective Cohort Study. Gastroenterol Res Pract. 2017;2017:4596176. doi: 10.1155/2017/4596176. Epub 2017 Feb 21. PMID 28316621
- [Background] Tempfer CB, Hartmann F, Hilal Z, Rezniczek GA. Intraperitoneal cisplatin and doxorubicin as maintenance chemotherapy for unresectable ovarian cancer: a case report. BMC Cancer. 2017 Jan 6;17(1):26. doi: 10.1186/s12885-016-3004-8. PMID 28061769
- [Background] Girshally R, Demtroder C, Albayrak N, Zieren J, Tempfer C, Reymond MA. Pressurized intraperitoneal aerosol chemotherapy (PIPAC) as a neoadjuvant therapy before cytoreductive surgery and hyperthermic intraperitoneal chemotherapy. World J Surg Oncol. 2016 Sep 27;14(1):253. doi: 10.1186/s12957-016-1008-0. PMID 27678344
- [Background] Graversen M, Pfeiffer P, Mortensen MB. [Treatment of peritoneal carcinomatosis with pressurized intraperitoneal aerosol chemotherapy]. Ugeskr Laeger. 2016 May 23;178(21):V11150928. Danish. PMID 27237925
- [Background] Robella M, Vaira M, De Simone M. Safety and feasibility of pressurized intraperitoneal aerosol chemotherapy (PIPAC) associated with systemic chemotherapy: an innovative approach to treat peritoneal carcinomatosis. World J Surg Oncol. 2016 Apr 29;14:128. doi: 10.1186/s12957-016-0892-7. PMID 27125996
- [Background] Tempfer CB, Rezniczek GA, Ende P, Solass W, Reymond MA. Pressurized Intraperitoneal Aerosol Chemotherapy with Cisplatin and Doxorubicin in Women with Peritoneal Carcinomatosis: A Cohort Study. Anticancer Res. 2015 Dec;35(12):6723-9. doi: 10.1055/s-0035-1560004. PMID 26637888
- [Background] Nadiradze G, Giger-Pabst U, Zieren J, Strumberg D, Solass W, Reymond MA. Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) with Low-Dose Cisplatin and Doxorubicin in Gastric Peritoneal Metastasis. J Gastrointest Surg. 2016 Feb;20(2):367-73. doi: 10.1007/s11605-015-2995-9. Epub 2015 Oct 28. PMID 26511950
- [Background] Demtroder C, Solass W, Zieren J, Strumberg D, Giger-Pabst U, Reymond MA. Pressurized intraperitoneal aerosol chemotherapy with oxaliplatin in colorectal peritoneal metastasis. Colorectal Dis. 2016 Apr;18(4):364-71. doi: 10.1111/codi.13130. PMID 26400556
- [Background] Hubner M, Teixeira H, Boussaha T, Cachemaille M, Lehmann K, Demartines N. [PIPAC--Pressurized intraperitoneal aerosol chemotherapy. A novel treatment for peritoneal carcinomatosis]. Rev Med Suisse. 2015 Jun 17;11(479):1325-30. French. PMID 26255492
- [Background] Odendahl K, Solass W, Demtroder C, Giger-Pabst U, Zieren J, Tempfer C, Reymond MA. Quality of life of patients with end-stage peritoneal metastasis treated with Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC). Eur J Surg Oncol. 2015 Oct;41(10):1379-85. doi: 10.1016/j.ejso.2015.06.001. Epub 2015 Jun 21. PMID 26138283
- [Background] Tempfer CB, Solass W, Buerkle B, Reymond MA. Pressurized intraperitoneal aerosol chemotherapy (PIPAC) with cisplatin and doxorubicin in a woman with pseudomyxoma peritonei: A case report. Gynecol Oncol Rep. 2014 Oct 18;10:32-5. doi: 10.1016/j.gore.2014.10.001. eCollection 2014 Dec. PMID 26076000
- [Background] Giger-Pabst U, Solass W, Buerkle B, Reymond MA, Tempfer CB. Low-dose pressurized intraperitoneal aerosol chemotherapy (PIPAC) as an alternative therapy for ovarian cancer in an octogenarian patient. Anticancer Res. 2015 Apr;35(4):2309-14. PMID 25862894
- [Background] Tempfer CB, Winnekendonk G, Solass W, Horvat R, Giger-Pabst U, Zieren J, Rezniczek GA, Reymond MA. Pressurized intraperitoneal aerosol chemotherapy in women with recurrent ovarian cancer: A phase 2 study. Gynecol Oncol. 2015 May;137(2):223-8. doi: 10.1016/j.ygyno.2015.02.009. Epub 2015 Feb 18. PMID 25701703
- [Background] Sabaila A, Fauconnier A, Huchon C. [Pressurized intraperitoneal aerosol chemotherapy (PIPAC): a new way of administration in peritoneal carcinomatosis of ovarian cancer]. Gynecol Obstet Fertil. 2015 Jan;43(1):66-7. doi: 10.1016/j.gyobfe.2014.11.012. Epub 2014 Dec 15. No abstract available. French. PMID 25523545
- [Background] Tempfer CB, Solass W, Reymond MA. Pressurized intraperitoneal chemotherapy (PIPAC) in women with gynecologic malignancies: a review. Wien Med Wochenschr. 2014 Dec;164(23-24):519-28. doi: 10.1007/s10354-014-0312-y. Epub 2014 Sep 24. PMID 25249025
- [Background] Tempfer CB, Celik I, Solass W, Buerkle B, Pabst UG, Zieren J, Strumberg D, Reymond MA. Activity of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) with cisplatin and doxorubicin in women with recurrent, platinum-resistant ovarian cancer: preliminary clinical experience. Gynecol Oncol. 2014 Feb;132(2):307-11. doi: 10.1016/j.ygyno.2013.11.022. Epub 2013 Nov 23. PMID 24275155
- [Background] Solass W, Kerb R, Murdter T, Giger-Pabst U, Strumberg D, Tempfer C, Zieren J, Schwab M, Reymond MA. Intraperitoneal chemotherapy of peritoneal carcinomatosis using pressurized aerosol as an alternative to liquid solution: first evidence for efficacy. Ann Surg Oncol. 2014 Feb;21(2):553-9. doi: 10.1245/s10434-013-3213-1. Epub 2013 Sep 5. PMID 24006094
- [Derived] Kurtz F, Struller F, Horvath P, Solass W, Bosmuller H, Konigsrainer A, Reymond MA. Feasibility, Safety, and Efficacy of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) for Peritoneal Metastasis: A Registry Study. Gastroenterol Res Pract. 2018 Oct 24;2018:2743985. doi: 10.1155/2018/2743985. eCollection 2018. PMID 30473706